CLINICAL TRIAL: NCT02246023
Title: Target-controlled Versus Manually-controlled Propofol Sedation in Flexible Bronchoscopy. A Randomized Non-inferiority Trial.
Brief Title: Fractionated Versus Target-controlled Propofol Administration in Bronchoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Franzen (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor-Investigator, Daniel Franzen, Dr. Daniel Franzen, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BronchoPropTCI; SNCTP000000706 (Registry Identifier: National study registration)
Record Dates: First submitted 2014-09-15; First posted 2014-09-22 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2015-06

CONDITIONS: Lung Cancer; Sarcoidosis; Interstitial Pneumonia
MeSH Terms: conditions — Lung Neoplasms; Sarcoidosis; Lung Diseases, Interstitial | interventions — Conscious Sedation; Blood Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fractionated propofol administration (Active Comparator): Flexible bronchoscopy in moderate sedation with fractionated propofol administrations: Patients receive an initial 20 mg of propofol, followed by a carefully titrated dose of10-20 mg propofol based on the clinical response.
  Continuous measurement of oxygen saturation Measurement of non-invasive blood pressure; Report of dose adjustments und cumulative propofol dosage; Recovery time after bronchoscopy
  Interventions: Device: Flexible bronchoscopy in moderate sedation; Device: Oxygen saturation; Device: Blood pressure; Device: Propofol dosage; Device: Recovery time after bronchoscopy
- Propofol-TCI (Experimental): Flexible bronchoscopy in moderate sedation with TCI propofol perfusor:
  Flexible bronchoscopy is started after reaching the initial targeted effect-site concentration (Ce) of 2.5 μg/mL using the Schnider pharmacokinetic model described elsewhere. Thereafter, Ce is adjusted by increments of 0.2 μg/mL depending on the clinical effect, in order to maintain the required level of sedation.
  Continuous measurement of oxygen saturation Measurement of non-invasive blood pressure; Report of dose adjustments und cumulative propofol dosage; Recovery time after bronchoscopy The propofol-TCI perfusor is an active infusion system for fluid management. In the study, the Perfusor® Space of B. Braun AG, Melsungen is used exclusively.
  Interventions: Device: Flexible bronchoscopy in moderate sedation; Device: Oxygen saturation; Device: Blood pressure; Device: Propofol dosage; Device: Recovery time after bronchoscopy

INTERVENTIONS:
Device: Flexible bronchoscopy in moderate sedation — Flexible bronchoscopy for diagnosis of lung cancer, sarcoidosis or interstitial pneumonia in moderate sedation with propofol;
Device: Oxygen saturation — Continuous measurement of oxygen saturation;
Device: Blood pressure — Measurement of non-invasive blood pressure every 3 minutes
Device: Propofol dosage — Report of dose adjustments und cumulative propofol dosage;
Device: Recovery time after bronchoscopy — Recovery time after bronchoscopy from removal of bronchoscope to eye opening/answer to verbal stimuli (whatever comes first)

SUMMARY:
After randomization, the subjects undergo flexible bronchoscopy either with fractionated propofol administration or with propofol-TCI. Measurement of blood pressure, heart rate, oxygen saturation, and oxygen requirement are measured continuously during the procedure and thereafter. Cumulative propofol dose, and induction, procedure, and recovery time are noted continuously during and after the procedure.

DETAILED DESCRIPTION:
In daily clinical praxis, propofol sedation is given manually in repeated doses (fractionated) by a specially-trained nurse in attendance of the bronchoscopist. But, fractionated propofol administration (FPA) may lead to oversedation and enhanced side effects (oxygen desaturation and arterial hypotension), as a stable plasma concentration of propofol is not maintainable. In contrast to FPA, continuous infusions of propofol are commonly used to induce and maintain long-term sedation in intensive care units and general anesthesia. Recently, continuous propofol infusion for sedation in bronchoscopy has been shown comparable to FPA in terms of safety and efficacy. Generally, infusion devices can be manually controlled (MCI) or target-controlled (TCI). In the latter, the physician sets a target blood concentration and the computerized infusion device makes the necessary changes to the infusion rate.

The objective of this study is to compare propofol TCI with FPA in flexible bronchoscopy concerning patient safety and sedation quality.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing a planned, ambulatory flexible bronchoscopy (for transbronchial lung biopsy or endobronchial ultrasound guided procedures) in moderate sedation, aged between 18 and 85 years

Exclusion Criteria:

* History of solid organ or bone marrow transplantation with the use of an immunosuppressive therapy
* HIV infection on anti-retroviral therapy
* Alcohol consumption more than two standard drinks per day
* Use of illicit drugs (heroin, opiates)
* Any contraindication to use propofol for sedation (e.g. allergy)
* Body mass index > 35 kg/m2
* Mental disorder preventing appropriate judgment concerning study participation
* Missing written patient's informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Mean arterial oxygen saturation | During bronchoscopy
  From induction of sedation until recovery (eye opening/answer to verbal stimuli), in average 45 minutes

SECONDARY OUTCOMES:
Number of occasions with recorded an oxygen saturation of < 90% | During bronchoscopy
  From induction of sedation until recovery (eye opening/answer to verbal stimuli), in average 45 minutes
Number of an oxygen desaturation of > 4% from baseline | During bronchoscopy
  From induction of sedation until recovery (eye opening/answer to verbal stimuli), in average 45 minutes
Number of occasions with a systolic blood pressure < 90 mmHg during bronchoscopy, maximum oxygen requirement, | During bronchoscopy
  From induction of sedation until recovery (eye opening/answer to verbal stimuli), in average 45 minutes
Frequency of dose adjustments | During bronchoscopy
  From induction of sedation until recovery (eye opening/answer to verbal stimuli), in average 45 minutes
Cumulative propofol dose | At end of bronchoscopy
  At time point when bronchoscope is removed (on average after 45 minutes)
Recovery time after bronchoscopy | During 2 hours after bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, MD, Principal Investigator — Division of Pulmonology
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland